CLINICAL TRIAL: NCT06284187
Title: Diagnosis Test of Real-time Polymerase Chain Reaction (RT-PCR) for Pulmonary Tuberculosis
Status: Completed | Type: Observational
Sponsor: Khon Kaen Hospital (Other Government)
Responsible Party: Principal Investigator, Kriengsak Vacharanukulkieti, Director of Hospital, Khon Kaen Hospital
Other Study IDs: KhonKaenH
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis; Pulmonary
Keywords: pulmonary tuberculosis; real-time PCR; diagnosis test
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND: Pulmonary tuberculosis remains the leading cause of morbidity and mortality in Thailand. The microbiological detection of TB is important because of early and correct diagnosis, drug resistance testing and ensures that the effective treatment can be achieved and in a timely manner. Mycobacterial culture is the gold standard diagnostic test. Currently, a real-time polymerase chain reaction (RT-PCR) assay, such as Allplex™ MTB/MDRe Detection, Seegene is commonly used.

OBJECTIVE: To evaluate the diagnosis value of the real-time multiplex PCR by using Allplex™ MTB/MDRe Detection kit to detect MTB from sputum specimens with a gold standard TB culture.

DETAILED DESCRIPTION:
A retrospective study design of adult patients (> 15 years) with suspected pulmonary M. tuberculosis infection was conducted from January 2023 until October 2023, at Khon Kaen Hospital. Sample size was 101 cases. Sensitivity, specificity, accuracy, negative predictive value (NPV), and positive predictive value (PPV) of Allplex™ MTB/MDRe Detection, each with its respective 95% confidence interval (95% CI) were analysed with compared to MTB culture as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspected pulmonary M. tuberculosis infection
* Aged 15 years and older

Exclusion Criteria:

* Children under 15 years old
* Non-tuberculous mycobacteria (NTM) detection

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: out patients clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with pulmonary TB by Allplex™ MTB/MDRe | From enrollment to the end of diagnosis at 1 week
  Laboratory parameter

CONTACTS AND LOCATIONS:
Overall Officials: Kriengsak Vacharanukulkieti, Medicine, Principal Investigator — Khon Kaen Hospital
Locations (1):
- Thananit Sangkomkamhang, Khon Kaen, Thailand